CLINICAL TRIAL: NCT01959334
Title: A Single Center, Randomized, Parallel Safety Study To Evaluate The Immunogenicity Of A Novel Glucagon Formulation Compared To Commercially Available Glucagon Administered By Intramuscular Injection In Adults With Type 1 OR Type 2 Diabetes
Brief Title: Evaluate the Immunogenicity of a Novel Glucagon Formulation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Locemia Solutions ULC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 16426; I8R-MC-IGBF (Other: Eli Lilly and Company); AMG105 (Other: Locemia Solutions ULC)
Record Dates: First submitted 2013-10-05; First posted 2013-10-10 (Estimated); Results first posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2016-04

CONDITIONS: Drug-specific Antibodies; Diabetes Mellitus
Keywords: Diabetes Mellitus; Hypoglycemia; Glucagon; Anti-glucagon Antibody; Immunogenicity
MeSH Terms: conditions — Diabetes Mellitus; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glucagon IM (Active Comparator): Glucagon dose of 1 milligram (mg) administered intramuscularly (IM).
  Interventions: Drug: Glucagon IM
- Nasal Glucagon (NG (Experimental): Nasal Glucagon (NG) doses of 3 mg administered intra-nasally.
  Interventions: Drug: Nasal Glucagon (NG)

INTERVENTIONS:
Drug: Nasal Glucagon (NG)
  Other Names: Nasal Glucagon; AMG504-1 Dry-Mist Intranasal Glucagon; LY900018
  Arms: Nasal Glucagon (NG
Drug: Glucagon IM
  Other Names: GlucaGen® HypoKit
  Arms: Glucagon IM

SUMMARY:
This study provides information on immunogenicity of Nasal Glucagon (AMG504-1) with regards to the potential development of treatment-emergent anti-glucagon antibodies.

DETAILED DESCRIPTION:
This study is a single center, randomized, laboratory-blinded, three periods, parallel design study.

The main objective of this study is to evaluate the immunogenicity of repeated single doses of glucagon following nasal and intramuscular (IM) administration in adults with Type 1 or Type 2 diabetes (T1D or T2D). The secondary objective is to evaluate the safety and tolerability of glucagon following NG and IM administration in adults with T1D or T2D.

A single dose of glucagon was administered in the morning after a 10-hour overnight fast, either by intranasal or intramuscular route, on 3 occasions. Each drug administration was separated by at least seven calendar days. Patients were randomized in a 2:1 ratio (NG:IMG) to receive NG or IMG at each of the 3 periods.

Blood samples were collected for measurement of anti-glucagon antibodies at screening visit, prior to dosing at Period 3, and at the post-study visit (approximately 4 weeks after the last glucagon administration).

ELIGIBILITY:
Inclusion Criteria:

1. Availability for the entire study period
2. Motivated volunteer and absence of intellectual problems likely to limit the validity of consent to participate in the study or the compliance with protocol requirements; ability to cooperate adequately; ability to understand and observe the instructions of the physician or designee
3. Male or female patient with a history of Type 1 or Type 2 diabetes of at least 2 years duration
4. A female volunteer must meet one of the following criteria:

   1. Participant is of childbearing potential and agrees to use one of the accepted contraceptive regimens throughout the entire duration of the study (from the screening visit until study completion). Additionally, if the participant is using systemic contraceptives, she must use an additional form of acceptable contraception. An acceptable method of contraception includes one of the following:

      * Abstinence from heterosexual intercourse
      * Systemic contraceptives (birth control pills, injectable/implant /insertable hormonal birth control products, transdermal patch)
      * Intrauterine device (with and without hormones)
      * Condom with spermicide

      or
   2. Participant is of non-childbearing potential, defined as surgically sterile (i.e. has undergone complete hysterectomy, bilateral oophorectomy, or tubal ligation) or in a menopausal state (at least 1 year without menses)
5. Volunteer aged of at least 18 years but not older than 70 years
6. Volunteer with a BMI greater than or equal to 18.50 and below 35.00 kg/m2
7. Light-, non- or ex-smokers. A light smoker is defined as someone smoking 10 cigarettes or less per day for at least 3 months before day 1 of this study. An ex- smoker is defined as someone who completely stopped smoking for at least 6 months before day 1 of this study
8. In good general health with no conditions that could influence the outcome of the trial, and in the judgment of the Investigator is a good candidate for the study based on review of available medical history, physical examination and clinical laboratory evaluations
9. Willingness to adhere to the protocol requirements as evidenced by the informed consent form (ICF) duly read, signed and dated by the volunteer

The informed consent form must be signed by all volunteers, prior to their participation in the study.

Exclusion Criteria:

1. Females who are pregnant, actively attempting to get pregnant, or are lactating
2. History of significant hypersensitivity to glucagon or any related products as well as severe hypersensitivity reactions (such as angioedema) to any drugs
3. Presence of significant gastrointestinal, liver or kidney disease, or any other conditions which in the judgment of the Investigator could interfere with the absorption, distribution, metabolism or excretion of drugs, or could potentiate or predispose to undesired effects
4. Suicidal tendency, history of or disposition to seizures, state of confusion, clinically relevant psychiatric diseases
5. Known presence of rare hereditary problems of galactose and /or lactose intolerance
6. Known presence or history of pheochromocytoma (i.e. adrenal gland tumor) or insulinoma (i.e. insulin secreting pancreas tumor)
7. Presence of clinically significant findings on nasal examination or bilateral anterior rhinoscopy, such as structural abnormalities, nasal polyps, marked septal deviation, nasal tumors
8. Nasal surgery in the previous 28 days before Day 1 of this study
9. Use of a systemic beta-blocker drug, indomethacin, warfarin or anticholinergic drugs in the previous 28 days before Day 1 of this study
10. Use of an immunomodulator medication (including steroids, glucocorticoids, tacrolimus, etc.) in the 28 days before day 1 of this study
11. Any other concomitant maintenance therapy that would influence the outcome of the trial or compromise the safety of the patient, at the discretion of the Investigator and the Sponsor, in the previous 28 days before day 1 of this study
12. Significant history of drug dependency or alcohol abuse (> 3 units of alcohol per day, intake of excessive alcohol, acute or chronic)
13. Any clinically significant illness in the previous 28 days before day 1 of this study
14. Any history of tuberculosis and/or prophylaxis for tuberculosis
15. Positive urine screening of alcohol and/or drugs of abuse
16. Females who are pregnant according to a positive pregnancy test
17. Concurrent participation or intention of participating in another clinical trial during this study
18. Volunteers who took an Investigational Product (in another clinical trial) or donated 50 mL or more of blood in the previous 28 days before day 1 of this study
19. Donation of 500 mL or more of blood (Canadian Blood Services, Hema-Quebec, clinical studies, etc.) in the previous 56 days before day 1 of this study

No participants will be allowed to enroll in this study more than once (i.e. if the study is conducted with more than 1 group).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2013-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Algorithme Pharma Inc., Laval, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Lilly provides access to the individual patient data from studies on approved medicines and indications as defined by the sponsor specific information on ClinicalStudyDataRequest.com.
  This access is provided in a timely fashion after the primary publication is accepted. Researchers need to have an approved research proposal submitted through ClinicalStudyDataRequest.com. Access to the data will be provided in a secure data sharing environment after signing a data sharing agreement.

RESULTS

PARTICIPANT FLOW:
Groups:
- Glucagon IM: Glucagon dose of 1 milligram (mg) administered intramuscularly as 3 doses separated by at least 7 days.
- Nasal Glucagon (NG): NG administered at 3 mg as 3 doses, separated by at least 7 days.
Period: First Dose
Arm/Group | Glucagon IM | Nasal Glucagon (NG)
Started | 26 | 49
Completed | 26 (Each Dosing Period separated by at least 7 calendar days.) | 49 (Each Dosing Period is separated by at least 7 calendar days.)
Not Completed | 0 | 0
Period: Second Dose
Arm/Group | Glucagon IM | Nasal Glucagon (NG)
Started | 26 | 49
Completed | 25 | 49
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Third Dose
Arm/Group | Glucagon IM | Nasal Glucagon (NG)
Started | 25 | 49
Completed | 25 | 48
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Glucagon IM: Glucagon dose of 1 mg administered intramuscularly as 3 doses separated by at least 7 days.
- Total: Total of all reporting groups
Arm/Group | Glucagon IM | Nasal Glucagon (NG) | Total
Number analyzed (Participants) | 26 | 49 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (12) | 43 (15) | 43 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 13 | 19
  Male | 20 | 36 | 56
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 24 | 44 | 68
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 26 | 49 | 75
BMI (Body Mass Index) [Mean (Standard Deviation); unit: kilogram per square metre (kg/m2)] | 27.08 (4.28) | 27.18 (3.93) | 27.15 (4.03)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-emergent Anti-Drug Antibody (ADA)
Description: Glucagon anti-drug antibodies (ADA) were assessed at baseline through study completion. Percentage of participants (Pts) with ADA=(number of Pts with treatment-emergent ADA/number of Pts assessed)*100. Treatment-Emergent ADA includes treatment-induced ADA and treatment boosted ADA. Treatment-induced is defined as participants with 'Not Detected' ADA at baseline (drug-naive) and at least one post-baseline ADA 'Detected' sample with a corresponding titer that is one 2-fold dilution higher than the MRD (minimal required dilution) of the assay. For the nasal glucagon Tier 1-3 ADA screening assay, the MRD is 1:20. Treatment-boosted is defined as Patient with ADA 'Detected' at baseline (drug-naive) and at least one post-baseline ADA 'Detected' sample with a corresponding titer that is at least (>or=) 4-fold higher than the baseline titer.
Time Frame: Baseline through study completion (up to 10 weeks)
Population: All enrolled participants who received at least 1 dose of study drug with an evaluable baseline ADA result and a post-baseline ADA result.
Measure: Number; unit: percentage of participants
Arm/Group | Glucagon IM | Nasal Glucagon (NG)
Number analyzed (Participants) | 26 | 49
percentage of participants | 0 | 2.0

2. Primary Outcome: Percentage of Participants With Neutralizing Antibodies
Time Frame: Baseline through study completion (up to 10 weeks)
Population: All enrolled participants who received at least 1 dose of study drug and either had baseline and at least 1 post-baseline evaluable samples or had no evaluable baseline and all negative post-baseline anti-drug antibody negative samples.
Measure: Number; unit: percentage of participants
Arm/Group | Glucagon IM | Nasal Glucagon (NG)
Number analyzed (Participants) | 26 | 49
percentage of participants | 0 | 0

3. Primary Outcome: Number of Participants With At Least One Adverse Event
Description: Safety parameters assessed included the occurrence of adverse events, the measurement of clinical laboratory parameters; vital signs, ECGs, physical examination, blood glucose, and examination of the injection site (following the IM administration). An AE was defined as any untoward medical occurrence in a clinical investigation subject administered the investigational product and which did not necessarily have a causal relationship with this treatment
  A summary of other nonserious AEs, and all SAE's, regardless of causality, is located in the Reported Adverse Events section.
Time Frame: First dose of study drug through the post-study completion (up to 10 weeks)
Population: Participants who received at least one dose of glucagon (IM or NG).
Measure: Count of Participants; unit: Participants
Arm/Group | Glucagon IM | Nasal Glucagon (NG)
Number analyzed (Participants) | 26 | 49
Participants | 21 | 49

ADVERSE EVENTS:
Time Frame: The period of observation of adverse events extended from time of the first dose of study drug until the post-study completion (up to 10 weeks).
Arm/Group | Glucagon IM | Nasal Glucagon (NG)
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/49
Other Adverse Events (participants affected / at risk) | 21/26 | 49/49
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glucagon IM (N=26) | Nasal Glucagon (NG) (N=49)
Headache (Nervous system disorders) | 3 (5) | 25 (38)
Somnolence (Nervous system disorders) | 4 (4) | 6 (6)
Dizziness (Nervous system disorders) | 3 (4) | 7 (10)
Dysgeusia (Nervous system disorders) | 0 (0) | 7 (12)
Parosmia (Nervous system disorders) | 0 (0) | 6 (6)
Tremor (Nervous system disorders) | 3 (3) | 3 (3)
Sinus headache (Nervous system disorders) | 0 (0) | 2 (3)
Lacrimation increased (Eye disorders) | 0 (0) | 48 (154)
Ocular hyperaemia (Eye disorders) | 1 (1) | 21 (30)
Eye pruritus (Eye disorders) | 0 (0) | 15 (19)
Eye irritation (Eye disorders) | 0 (0) | 3 (4)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 20 (53)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 21 (67)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 20 (28)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 12 (17)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 7 (8)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 7 (8)
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Injection site pain (General disorders) | 6 (8) | 0 (0)
Fatigue (General disorders) | 3 (3) | 3 (3)
Feeling hot (General disorders) | 1 (1) | 4 (4)
Injection site anaesthesia (General disorders) | 3 (4) | 0 (0)
Injection site reaction (General disorders) | 3 (3) | 0 (0)
Injection site discomfort (General disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 13 (30)
Vomiting (Gastrointestinal disorders) | 2 (4) | 9 (22)
Hot flush (Vascular disorders) | 3 (3) | 5 (6)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 3 (6)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (3)
Ear pruritus (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Eye Pain (Eye disorders) | 0 (0) | 2 (2)
Ocular discomfort (Eye disorders) | 0 (0) | 3 (3)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abnormal faeces (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Administration site reaction (General disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 2 (3)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Feeling cold (General disorders) | 1 (1) | 1 (1)
Injection site hypoaesthesia (General disorders) | 2 (3) | 0 (0)
Injection site paraesthesia (General disorders) | 1 (1) | 0 (0)
Injection site warmth (General disorders) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 2 (3)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (4)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (2)
Administration related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood glucose decreased (Investigations) | 1 (1) | 0 (0)
Blood sodium decreased (Investigations) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Head discomfort (Nervous system disorders) | 0 (0) | 5 (5)
Pallor (Vascular disorders) | 0 (0) | 2 (3)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal pruritus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 17 (25)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
This study was conducted by a Contract Research Organization. The Sponsor is and shall remain owner of all data pertaining to and/or resulting from the Study as well as all rights on intellectual property and patents arising from the said Study. Confidential Information may not be disclosed to any third party without the other party's prior written consent (except to the relevant authorities, providing the confidentiality is maintained).